CLINICAL TRIAL: NCT03710538
Title: The Effect of a Pre-meal Snack and/or Exercise on Post-prandial Glycemic Excursions in Adults With Cystic Fibrosis
Acronym: SNACK_CF
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Institut de Recherches Cliniques de Montreal (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Single | Purpose: Treatment
Other Study IDs: SNACK_CF
Record Dates: First submitted 2018-06-20; First posted 2018-10-18 (Actual); Last update posted 2023-04-25 (Actual); Status verified 2023-04

CONDITIONS: Cystic Fibrosis
Keywords: glycemia
MeSH Terms: conditions — Cystic Fibrosis | interventions — Exercise

STUDY DESIGN:
Intervention Model Description: 1. Consumption of 200ml of water (flavored) + breakfast of 90g of carbohydrates (CHO) for men and 80g for women; Sedentary activities throughout the study [condition control]
  2. Consumption of 200ml of soy beverage + 90g of carbohydrate (CHO) breakfast for men and 80g for women; Sedentary activities throughout the study [snack effect on PPG excursion]
  3. Consumption of 200ml of water (flavored) + breakfast of 90g of carbohydrates (CHO) for men and 80g for women + physical activity practice (3min walk at 60% VO2max every 30 minutes, x5); [exercise effect on the PPG excursion]
  4. Consumption of 200ml of soy beverage + breakfast of 90g of carbohydrate (CHO) breakfast for men and 80g for women + physical activity practice (3min walk at 60% VO2max every 30 minutes, x5). [Combined snack and exercise effect on the PPG excursion]
Who Masked: Participant
Masking Description: snack beverage or flavored placebo will be not recognizable
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- [Placebo + Sedentary] (No Intervention): 1) Consumption of 200ml of water (flavored) + breakfast of 90g of carbohydrates (CHO) for men and 80g for women; Sedentary activities throughout the study
- [Snack effect + Sedentary] (Experimental): 2) Consumption of 200ml of soy beverage + 90g of carbohydrate (CHO) breakfast for men and 80g for women; Sedentary activities throughout the study
  Interventions: Dietary Supplement: Snack beverage
- [Placebo + Exercise] (Experimental): 3) Consumption of 200ml of water (flavored) + breakfast of 90g of carbohydrates (CHO) for men and 80g for women + physical activity practice (3min walk at 60% VO2max every 30 minutes, x5);
  Interventions: Behavioral: Exercise
- [Snack + Exercise] (Experimental): 4) Consumption of 200ml of soy beverage + breakfast of 90g of carbohydrate (CHO) breakfast for men and 80g for women + physical activity practice (3min walk at 60% VO2max every 30 minutes, x5).
  Interventions: Dietary Supplement: Snack beverage; Behavioral: Exercise

INTERVENTIONS:
Dietary Supplement: Snack beverage — Consumption of a 200ml of soy beverage (100Kcal, 11g CHO, 6g proteins, 4g fat)
  Arms: [Snack + Exercise]; [Snack effect + Sedentary]
Behavioral: Exercise — 3min walk at 60% VO2max every 30 minutes,(x5)
  Arms: [Placebo + Exercise]; [Snack + Exercise]

SUMMARY:
The investigators aim to test the feasibility and effectiveness of a pre-meal snack to reduce the postprandial glycemia (PPG) excursion after a breakfast consumption in adult patients with cystic fibrosis (CF). The investigators also want to investigate the impact of a postprandial exercise to reduce the PPG excursion. An improvement in PPG excursions can improve the condition of CF patients primarily by delaying the onset of cystic fibrosis related diabetes (CFRD) and / or by reducing the risk of lung function loss.

DETAILED DESCRIPTION:
The investigators are proposing a randomized pilot study to explore the impact of a soy beverage of carbohydrates and protein early in the morning, to stimulate and initiate secretion of Insulin to reduce PPG excursions of the following a lunch in adult patients with CF. Investigators will also study the impact of a post meal exercise on the PPG excursion. Fourteen participants will be included and will each perform a 4-hour intervention in cross over design according to those 4 following experimental conditions:

1. Consumption of 200ml of water (flavored) + breakfast of 90g of carbohydrates (CHO) for men and 80g for women; Sedentary activities throughout the study [condition control]
2. Consumption of 200ml of soy beverage + 90g of carbohydrate (CHO) breakfast for men and 80g for women; Sedentary activities throughout the study [snack effect on PPG excursion]
3. Consumption of 200ml of water (flavored) + breakfast of 90g of carbohydrates (CHO) for men and 80g for women + physical activity practice (3min walk at 60% VO2max every 30 minutes, x5); [exercise effect on the PPG excursion]
4. Consumption of 200ml of soy beverage + breakfast of 90g of carbohydrate (CHO) breakfast for men and 80g for women + physical activity practice (3min walk at 60% VO2max every 30 minutes, x5). [Combined snack and exercise effect on the PPG excursion] Main result: plasma glucose area under the curve. The underlying mechanisms, insulin, incretin hormones (GLP-1 and GIP), acceptability and side effects (mealtime hyperglycaemia) should also be measured. At the end of this pilot project, the investigators will have established a pre-meal snack and/ or postprandial exercise have a positive impact on PPG.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of cystic fibrosis,
* Be over 18 years old.

Exclusion Criteria:

* Pharmacological treatment for cystic fibrosis related diabetes.
* Signs of secondary infection: the test will be practiced at least 1 month after the end of infection treatment
* People with severe gastrointestinal illness (Crohn's disease, celiac disease and a recent history (<1 year) of bowel obstruction).
* Allergy to one of the ingredients of the menu (example: celiac disease)
* According to the judgment of the investigator, medications or conditions that could interfere with glucose metabolism (eg: oral steroids)
* Pregnancy in progress
* Corrector or potentiator prescribed whose dose is not stable the last 2 months.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 14 (Actual)
Dates: Start 2019-04-01 (Actual); Primary Completion 2022-05-26 (Actual); Study Completion 2022-12-31 (Actual)

PRIMARY OUTCOMES:
Total area under the curve for plasma glucose | Overall study period (4 hours)

SECONDARY OUTCOMES:
Area under the curve for plasma glucose | From start of study to breakfast time (1 hour)
Area under the curve for plasma glucose | From time of breakfast to the end of the study (3 hours)
Total area under the curve for insulin | Overall study period (4 hours)
Area under the curve for insulin | From start of study to breakfast time (1 hour)
Area under the curve for insulin | From breakfast time to the end of the study (3 hours)
Mean plasma glucose | Overall study period (4 hours)
Mean insulin | Overall study period (4 hours)
Percentage of time with plasma glucose concentration above 8.0 mmol/L | Overall study period (4 hours)
Percentage of time with plasma glucose concentration above 10.0 mmol/L | Overall study period (4 hours)
Percentage of time with plasma glucose concentration above 11.0 mmol/L | Overall study period (4 hours)
Percentage of time with plasma glucose concentration below 4.0 mmol/L | Overall study period (4 hours)
Post-breakfast peak plasma glucose | 1 hour after breakfast

CONTACTS AND LOCATIONS:
Overall Officials: Rémi Rabasa-Lhoret, MD, PhD, Principal Investigator — IRCM
Locations (1):
- Institut de Recherches Cliniques de Montréal (IRCM), Montreal, Quebec, Canada

IPD SHARING:
Plan to Share IPD: No